CLINICAL TRIAL: NCT00733369
Title: A Prospective, Single Blinded, Multi-centre Randomised Controlled Trial Comparing the Post Operative Range of Motion of the P.F.C. Sigma RP-F Knee With the P.F.C. Sigma RP Knee in Primary Total Knee Arthroplasty.
Brief Title: A Study to Compare the Press Fit Condylar (P.F.C.) Sigma Rotating-platform High-flexion (RP-F) Versus the Press Fit Condylar (P.F.C.) Sigma Rotating-platform (RP) Knee Implants
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was closed for the reason of slow recruitment with only 16% of the target subjects recruited over a 29 month period.
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT 06/03
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Knee Osteoarthritis
Keywords: Arthroplasty; Replacement; Knee; PFC Sigma RPF; PFC Sigma RP
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PFC Sigma RP-F (Other): 125 patients to be allocated to this arm according to blinding envelopes
  Interventions: Device: PFC Sigma RP-F
- PFC Sigma RP (Active Comparator): 125 patients to be allocated to this arm according to blinding envelopes
  Interventions: Device: PFC Sigma RP

INTERVENTIONS:
Device: PFC Sigma RP-F — An orthopaedic implant for total knee replacement with a high flexion rotating platform bearing
  Arms: PFC Sigma RP-F
Device: PFC Sigma RP — An orthopaedic implant for total knee replacement with a standard flexion rotating platform bearing
  Arms: PFC Sigma RP

SUMMARY:
The main objective of this study is to determine if the P.F.C. Sigma RP-F Knee delivers a greater post-operative range of motion (ROM) compared with the P.F.C. Sigma RP Knee in primary TKA.

The secondary objectives of this investigation are to evaluate the clinical and patient outcomes and survivorship associated with the DePuy P.F.C. Sigma RP-F and RP Posterior Stabilised (PS) Knee over 5 years.

DETAILED DESCRIPTION:
Primary Outcome: Change from pre-operative range of motion at 1 year between patients receiving P.F.C. Sigma RP vs P.F.C. Sigma RP-F

Secondary endpoints: Comparative evaluation of any post-operative variation between subjects receiving primary TKA with either of the above devices in terms of Knee and Osteoarthritis Scores (KOOS), American Knee Society Score (AKS), EQ-5D Score and Oxford Knee Score (OKS)

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 45 and 75 years inclusive.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Subjects who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.
* Subjects who present with osteoarthritis that in the opinion of the clinical investigator requires a primary total knee arthroplasty.
* Subjects who in the opinion of the Clinical Investigator are considered to be suitable for treatment with either the P.F.C Sigma RP-F or the P.F.C Sigma RP knee, according to the indications specified in the package insert leaflet.
* Subjects who have authorised the transfer of his/her pseudonymised information to DePuy.

Exclusion Criteria:

* Subjects who, in the opinion of the Clinical Investigator, have an existing condition that would compromise their participation and follow-up in this clinical investigation.
* Female subjects who are pregnant or lactating.
* Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have participated in a clinical investigation with an investigational product in the last month( 30 days).
* Subjects who are currently involved in any injury litigation claims.
* Subjects with a known history of poor compliance to medical treatment.
* Subjects who have previously had an osteotomy or significant surgery in the affected knee.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-11; Primary Completion 2010-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Hospital Clinic i Provincial de Barcelona, Barcelona, Spain
- Arrowe Park Hospital, Metropolitan Borough of Wirral, Mersyside, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 sites enrolled 106 knees in 98 subjects who were then randomized into 2 groups, 50 into the PFC Sigma RP-F group and 56 into the PFC Sigma RP group.
Pre-assignment Details: Study protocol was designed and executed on using 'knees' as study units.
Groups:
- PFC Sigma RP-F: PFC Sigma RP-F : An orthopaedic implant for total knee replacement with a high flexion rotating platform bearing
- PFC Sigma RP: PFC Sigma RP : An orthopaedic implant for total knee replacement with a standard flexion rotating platform bearing
Period: Overall Study
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Started | 50 | 56
Completed | 40 | 47
Not Completed | 10 | 9
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 4 | 4
Not completed — Protocol Violation | 4 | 4

BASELINE CHARACTERISTICS:
Population: Study protocol was designed and executed on using 'knees' as study units. Out of 106 enrolled knees, 11 knees were removed from analysis for following reasons: 8 protocol violations [bilaterals accrued at site bilaterals not allowed; used 1st knee operated upon] (4 inv, 4 control); 2 ltfu (1 inv, 1 control); 1 missing outcome (1 inv, 0 control).
Groups:
- Total: Total of all reporting groups
Arm/Group | PFC Sigma RP-F | PFC Sigma RP | Total
Number analyzed (Participants) | 50 | 56 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (7.2) | 66.3 (6.4) | 65.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 42 | 72
  Male | 20 | 14 | 34
Region of Enrollment [Number; unit: participants]
  Spain | 48 | 52 | 100
  United Kingdom | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-op to 1 Year Range of Motion.
Description: Range of motion is knee flexion (how far the patient can bend their knee) minus knee extension (how far the patient can straighten their knee). The result of this subtraction is the range of motion (bending and straightening) for that knee.
Time Frame: 1 year
Population: 106 enrolled knees, 11 of which excluded from the analysis due to:{0 Deaths + 8 Protocol Violations(bilaterals accrued at site where bilateral not allowed, used first knee operated upon: 4 investigational &4 control) + 2 lost to follow up (1 Inv & 1 Contr) + 1 missing outcome (1 Inv & 0 Contr)}
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 51
Number analyzed (Number of Knees) | 44 | 51
Degrees | 13.11 (14.89) | 10.71 (14.38)

2. Secondary Outcome: To Compare the Change in KOOS Pain Score From Pre-Op to 3 to 6 Months Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: The Knee injury and Osteoarthritis Outcome Score (KOOS) is a patient reported outcome that evaluates the short and long-term symptoms and function in subjects with knee injury and osteoarthritis. It consists of 5 separately scored subscales - Pain, Symptoms, Function in daily living (ADL), Function in Sport and Recreation, and knee-related Quality of Life (QOL) - ranging from 0 to 100 point score (where 100 indicates the best outcome).
Time Frame: 3-6 months
Population: 106 Enrolled knees, 11 of which excluded from analysis due to:{0 Deaths+8 Protocol Violations(4Inv & 4Contr)+1 Lost to follow up(1Inv & 0Contr)+2 Missing outcome(1Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 51
Number analyzed (Number of Knees) | 44 | 51
Points | 39.7 (21.7) | 46.5 (18.0)

3. Secondary Outcome: To Compare the Change in KOOS Pain Score From Pre-Op to 1 Year Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 1 year
Population: 106 enrolled knees, 11 of which were excluded from analysis due to:{0 Deaths + 8 Protocol Violations (Bilaterals accrued at site where bilaterals are not allowed, used 1st knee operated upon: 4 investigational&4control)+ 2 lost to follow up (1 Inv, 1 Contr)+ 1 missing outcome (0Inv, 1 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 50
Number analyzed (Number of Knees) | 45 | 50
Points | 45.0 (20.5) | 48.9 (19.4)

4. Secondary Outcome: To Compare the Change in KOOS Pain Score From Pre-Op to 2 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 2 years
Population: 106 enrolled knees, 15 of which excluded from analysis due to:{0 Deaths + 8 Protocol Violation (4 Inv, 4 Contr) + 4 Revisions (1 Inv, 3 Contr) + 3 Lost to follow up (2 Inv, 1 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 48
Number analyzed (Number of Knees) | 43 | 48
Points | 43.3 (21.3) | 47.8 (20.1)

5. Secondary Outcome: To Compare the Change in KOOS Pain Score From Pre-Op to 5 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 5 years
Population: This study has been terminated early, therefore the 5 year data was not collected.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

6. Secondary Outcome: To Compare the Change in KOOS Symptoms Score From Pre-Op to 3 to 6 Months Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 3-6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 51
Number analyzed (Number of Knees) | 44 | 51
Points | 23.1 (18.4) | 32.4 (21.1)

7. Secondary Outcome: To Compare the Change in KOOS Symptoms Score From Pre-Op to 1 Year Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 1 year
Population: 106 enrolled knees, 11 of which excluded from the analysis due to:{0 Deaths+8 Protocol Violations (4 Inv & 4 Contr)+ 2 Lost to follow up (1 Inv & 1 Contr) + 1 Missing outcome (0 Inv & 1 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 50
Number analyzed (Number of Knees) | 45 | 50
Points | 29.8 (21.7) | 30.5 (22.1)

8. Secondary Outcome: To Compare the Change in KOOS Symptoms Score From Pre-Op to 2 Years Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 2 years
Population: 106 enrolled knees, 15 of which excluded from the analysis due to:{0 Deaths+8 Protocol Violations (4 Inv & 4 Contr)+ 4 Revisions (1 Inv & 1 Contr)+ 3 Lost to follow up (2 Inv & 1 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 48
Number analyzed (Number of Knees) | 43 | 48
Points | 30.5 (20.9) | 33.5 (25.0)

9. Secondary Outcome: To Compare the Change in KOOS Symptoms Score From Pre-Op to 5 Years Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 5 years
Population: This study was terminated early due to a slow recruitment rate. 5 year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

10. Secondary Outcome: To Compare the Change in KOOS ADL (Activities of Daily Living) Score From Pre-Op to 3 to 6 Months Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 3-6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 51
Number analyzed (Number of Knees) | 44 | 51
Points | 36.0 (18.7) | 43.7 (20.1)

11. Secondary Outcome: To Compare the Change in KOOS ADL (Activities of Daily Living) Score From Pre-Op to 1 Year Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 1 year
Population: 106 enrolled knees, 11 of which excluded from analysis due to:{0 Deaths + 8 Protocol Violations (4 Inv & 4 Contr)+ 2 Lost to follow up (1 Inv & 1 Contr) + 1 Missing outcome (0 Inv & 1 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 50
Number analyzed (Number of Knees) | 45 | 50
Points | 41.5 (18.5) | 44.0 (23.0)

12. Secondary Outcome: To Compare the Change in KOOS ADL (Activities of Daily Living) Score From Pre-Op to 2 Years Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 2 years
Population: 106 enrolled knees, 15 of which excluded from the analysis due to:{0 Deaths+8 Protocol Violations (4 Inv & 4 Contr)+ 4 Revisions (1 Inv & 3 Contr) + 3 Lost to follow up (2 Inv & 1 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 48
Number analyzed (Number of Knees) | 43 | 48
Points | 39.6 (18.7) | 42.5 (23.5)

13. Secondary Outcome: To Compare the Change in KOOS ADL (Activities of Daily Living) Score From Pre-Op to 5 Years Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 5 years
Population: Study terminated early due to a slow recruitment rate.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

14. Secondary Outcome: To Compare the Change in KOOS SPORTS and RECREATION Score From Pre-Op to 3 to 6 Months Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 3-6 months
Population: 106 knees enrolled, 11 of which excluded from analysis due to: {0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 1 Lost to follow up (1Inv & 0Contr) + 2 Missing outcome (1Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 51
Number analyzed (Number of Knees) | 44 | 51
Points | 14.4 (22.3) | 17.4 (24.7)

15. Secondary Outcome: To Compare the Change in KOOS SPORTS and RECREATION Score From Pre-Op to 1 Year Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 1 year
Population: 106 enrolled knees, 13 of which excluded from analysis due to:{0 Deaths+8 Protocol Violations (4 Inv & 4 Contr)+ 2 Lost to follow up (1 Inv & 1 Contr) + 3 Missing outcome (0 Inv & 3 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 48
Number analyzed (Number of Knees) | 45 | 48
Points | 35.4 (27.7) | 33.5 (25.1)

16. Secondary Outcome: To Compare the Change in KOOS SPORTS and RECREATION Score From Pre-Op to 2 Years Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 2 years
Population: 106 enrolled knees, 16 of which excluded from analysis due to:{0 Deaths+8 Protocol Violations (4 Inv & 4 Contr)+ 4 Revisions (1 Inv & 3 Contr) + 3 Lost to follow up (2 Inv & 1 Contr) + 1 Missing outcome (1 Inv & 0 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 42 | 48
Number analyzed (Number of Knees) | 42 | 48
Points | 36.6 (27.8) | 37.8 (25.3)

17. Secondary Outcome: To Compare the Change in KOOS SPORTS and RECREATION Score From Pre-Op to 5 Years Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 5 years
Population: Study terminated early due to slow recruitment rate, 5 year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

18. Secondary Outcome: To Compare the Change in KOOS QOL (Quality of Life) Score From Pre-Op to 3 to 6 Months Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 3-6 months
Population: 106 knees enrolled, 11 of which excluded from analysis due to:{0 deaths + 8 Protocol Violations + 1 Lost to follow up (1Inv & 0Contr) + 2 Missing outcome (1Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 51
Number analyzed (Number of Knees) | 44 | 51
Points | 42.2 (26.7) | 48.0 (26.2)

19. Secondary Outcome: To Compare the Change in KOOS QOL (Quality of Life) Score From Pre-Op to 1 Year Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 1 year
Population: 106 enrolled knees, 13 of which excluded from the analysis due to:{0 Deaths+ 8 Protocol Violations (4 Inv & 4 Contr)+ 2 Lost to follow up (1 Inv & 1 Contr) + 3 Missing outcome (0 Inv & 3 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 48
Number analyzed (Number of Knees) | 45 | 48
Points | 49.0 (29.0) | 51.7 (27.7)

20. Secondary Outcome: To Compare the Change in KOOS QOL (Quality of Life) Score From Pre-Op to 2 Years Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 2 years
Population: 106 knees enrolled, 16 of which excluded from analysis due to: {0 Deaths + 8 Protocol Violations (4 Inv & 4 Contr) + 4 Revisions (1 Inv & 3 Contr) + 3 Lost to follow up (2 Inv & 1 Contr) + 1 Missing outcome (1 Inv & 0 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 42 | 48
Number analyzed (Number of Knees) | 42 | 48
Points | 44.3 (31.6) | 50.8 (23.6)

21. Secondary Outcome: To Compare the Change in KOOS QOL (Quality of Life) Score From Pre-Op to 5 Years Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 2
Time Frame: 5 years
Population: Study terminated early due to slow recruitment rate. 5 Year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

22. Secondary Outcome: To Compare the Change in American Knee Society (AKS) Knee Score From Pre-Op to 3 to 6 Months Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: American Knee Society (AKS) knee score is a 0-100 point score (where 100 indicates excellent knee condition) that evaluates the affected knee. The knee score is composed of Pain, Range of Motion, and Stability.
Time Frame: 3 - 6 months
Population: 106 knees enrolled, 10 of which were excluded from analysis due to:{0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 1 Lost to follow up (1Inv & 0Contr) + 1 Missing outcome (1Inv & 0Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 52
Number analyzed (Number of Knees) | 44 | 52
Points | 36.3 (17.9) | 39.1 (15.7)

23. Secondary Outcome: To Compare the Change in American Knee Society (AKS) Knee Score From Pre-Op to 1 Year Post Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 22
Time Frame: 1 year
Population: 106 enrolled knees, 11 knees excluded from analysis due to: {0 Deaths + 8 Protocol Violations (4 Inv, 4 Contr) + 2 lost to follow up (1 Inv, 1 Contr) + 1 missing outcome (1 Inv, 0 Contr) }
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 51
Number analyzed (Number of Knees) | 44 | 51
Points | 40.0 (17.6) | 38.9 (17.2)

24. Secondary Outcome: To Compare the Change in American Knee Society (AKS) Knee Score From Pre-Op to 2 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 22
Time Frame: 2 years
Population: 106 enrolled knees, 18 knees excluded from analysis due to: {0 Deaths + 8 Protocol Violations (4 Inv, 4 Contr) + 4 revisions (1 Inv, 1 Contr) + 3 Lost to follow up (2 Inv, 1 Contr) + 3 missing outcome (0 Inv, 3 Cntr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 45
Number analyzed (Number of Knees) | 43 | 45
Points | 37.3 (20.6) | 36.8 (19.6)

25. Secondary Outcome: To Compare the Change in American Knee Society (AKS) Knee Score From Pre-Op to 5 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 22
Time Frame: 5 years
Population: Study terminated early due to a slow recruitment rate. 5 year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

26. Secondary Outcome: To Compare the Change in American Knee Society (AKS) Function Score From Pre-Op to 3 to 6 Months Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: American Knee Society (AKS) function score is a 0-100 point score (where 100 indicates excellent knee function) that evaluates the affected knee.
Time Frame: 3 - 6 months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 52
Number analyzed (Number of Knees) | 44 | 52
Points | 25.0 (19.6) | 28.9 (17.3)

27. Secondary Outcome: To Compare the Change in American Knee Society (AKS) Function Score From Pre-Op to 1 Year Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 26
Time Frame: 1 year
Population: 106 knees enrolled, 11 of which were excluded from analysis due to:{0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 2 Lost to follow up (1Inv & 1Contr) + 1 Missing outcome (1Inv & 0Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 51
Number analyzed (Number of Knees) | 44 | 51
Points | 30.5 (19.3) | 30.1 (19.9)

28. Secondary Outcome: To Compare the Change in American Knee Society (AKS) Function Score From Pre-Op to 2 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 26
Time Frame: 2 years
Population: 106 knees enrolled, 16 of which were excluded from analysis due to:{0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 4 Revisions (1Inv & 3Contr) + 3 Lost to follow up (2Inv & 1Contr) + 1 Missing outcome (0Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 47
Number analyzed (Number of Knees) | 43 | 47
Points | 24.9 (18.4) | 26.5 (18.1)

29. Secondary Outcome: To Compare the Change in American Knee Society (AKS) Function Score From Pre-Op to 5 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 26
Time Frame: 5 years
Population: Study terminated early due to a slow recruitment rate. 5 Year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

30. Secondary Outcome: To Compare the Change in Oxford Knee Score (OKS) From Pre-Op to 3 to 6 Months Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: The Oxford Knee Score (OKS) is a 12 to 60 point patient reported outcome (PRO) score (where 12 indicates the best outcome) that evaluates the affected knee. The total score is composed of Pain and Function.
Time Frame: 3 - 6 months
Population: 106 knees enrolled, 10 of which were excluded from analysis due to:{0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 1 Lost to follow up (1Inv & 0Contr) + 1 Missing outcome (0Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 51
Number analyzed (Number of Knees) | 45 | 51
Points | -14.4 (8.8) | -18.0 (8.7)

31. Secondary Outcome: To Compare the Change in Oxford Knee Score (OKS) From Pre-Op to 1 Year Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 30
Time Frame: 1 year
Population: 106 knees enrolled, 12 of which were excluded from analysis due to:{0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 2 Lost to follow up (1Inv & 1Contr) + 2 Missing outcome (1Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 44 | 50
Number analyzed (Number of Knees) | 44 | 50
Points | -18.7 (8.6) | -19.4 (8.7)

32. Secondary Outcome: To Compare the Change in Oxford Knee Score (OKS) From Pre-Op to 2 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 30
Time Frame: 2 years
Population: 106 knees enrolled, 17 of which were excluded from analysis due to:{0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 4 Revisions (1Inv & 3Contr) + 3 Lost to follow up (2Inv & 1Contr) + 2 Missing outcome (0Inv & 2Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 46
Number analyzed (Number of Knees) | 43 | 46
Points | -17.3 (9.7) | -19.1 (9.6)

33. Secondary Outcome: To Compare the Change in Oxford Knee Score (OKS) From Pre-Op to 5 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 30
Time Frame: 5 years
Population: Study terminated early due to a slow recruitment rate. 5 Year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

34. Secondary Outcome: To Compare the Change in EQ-5D3L MOBILITY Score From Pre-Op to 3 to 6 Months Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: EQ-5D3L is a patient reported standardized instrument used to measure health that comprises of 5 descriptive dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; and 1 visual analog scale (VAS) that measures health. The descriptive dimensions each have 3 levels: no problems (scored as 1), some problems (scored as 2), and extreme problems (scored as 3); whereas the VAS measure ranges from 0 to 100 where 100 is the best imaginable health state.
Time Frame: 3 - 6 months
Population: 106 knees enrolled, 9 of which were excluded from analysis due to:{0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 1 Lost to follow up (1Inv & 0Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 52
Number analyzed (Number of Knees) | 45 | 52
Points | -0.58 (0.62) | -0.58 (0.57)

35. Secondary Outcome: To Compare the Change in EQ-5D3L MOBILITY Score From Pre-Op to 1 Year Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 1 year
Population: 106 knees enrolled, 11 of which were excluded from analysis due to:{0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 2 Lost to follow up (1Inv & 1Contr) + 1 Missing outcome (0Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 50
Number analyzed (Number of Knees) | 45 | 50
Points | -0.62 (0.58) | -0.50 (0.58)

36. Secondary Outcome: To Compare the Change in EQ-5D3L MOBILITY Score From Pre-Op to 2 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 2 years
Population: 106 knees enrolled, 15 of which were excluded from analysis due to:{0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 4 Revisions (1Inv & 3Contr) + 3 Lost to follow up (2Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 48
Number analyzed (Number of Knees) | 43 | 48
Points | -0.58 (0.63) | -0.48 (0.58)

37. Secondary Outcome: To Compare the Change in EQ-5D3L MOBILITY Score From Pre-Op to 5 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 5 years
Population: Study terminated early to slow recruitment rate. 5 Year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

38. Secondary Outcome: To Compare the Change in EQ-5D3L Self-Care Score From Pre-Op to 3 to 6 Months Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 3 - 6 months
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 52
Number analyzed (Number of Knees) | 45 | 52
Points | -0.04 (0.56) | -0.19 (0.56)

39. Secondary Outcome: To Compare the Change in EQ-5D3L Self-Care Score From Pre-Op to 1 Year Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 1 year
Population: 106 enrolled knees, 11 of which excluded from analysis due to: {0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 2 Lost to follow up (1 Inv & 1 Contr) + 1 Missing outcome ( 0 Inv & 1 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 50
Number analyzed (Number of Knees) | 45 | 50
Points | -0.11 (0.49) | -0.22 (0.58)

40. Secondary Outcome: To Compare the Change in EQ-5D3L Self-Care Score From Pre-Op to 2 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 2 years
Population: 106 enrolled knees, 15 of which excluded from analysis due to: {0 Deaths + 8 Protocol Violations (4Inv & 4Contr) + 4 Revisions (1 Inv & 3 Contr) + 3 Lost to follow up (2 Inv & 1 Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 48
Number analyzed (Number of Knees) | 43 | 48
Points | -0.07 (0.51) | -0.15 (0.55)

41. Secondary Outcome: To Compare the Change in EQ-5D3L Self-Care Score From Pre-Op to 5 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 5 years
Population: Study terminated early due to slow recruitment rate. 5 Year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

42. Secondary Outcome: To Compare the Change in EQ-5D3L Usual Activities Score From Pre-Op to 3 to 6 Months Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 3 - 6 months
Population: 106 knees enrolled, 9 of which excluded from analysis due to:{0Deaths + 8 Protocol Violations (4Inv & 4 Contr) + 1 Lost to follow up (1Inv & 0Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 52
Number analyzed (Number of Knees) | 45 | 52
Points | -0.40 (0.65) | -0.50 (0.58)

43. Secondary Outcome: To Compare the Change in EQ-5D3L Usual Activities Score From Pre-Op to 1 Year Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 1 year
Population: 106 knees enrolled, 11 of which excluded from analysis due to:{0Deaths + 8 Protocol Violations (4Inv & 4 Contr) + 2 Lost to follow up (1Inv & 1Contr) + 1 Missing outcome (0Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 50
Number analyzed (Number of Knees) | 45 | 50
Points | -0.53 (0.63) | -0.48 (0.61)

44. Secondary Outcome: To Compare the Change in EQ-5D3L Usual Activities Score From Pre-Op to 2 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 2 years
Population: 106 knees enrolled, 15 of which excluded from analysis due to:{0Deaths + 8 Protocol Violations (4Inv & 4 Contr) + 4 Revisions (1Inv & 3Contr) + 3 Lost to follow up (2Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 48
Number analyzed (Number of Knees) | 43 | 48
Points | -0.42 (0.59) | -0.44 (0.58)

45. Secondary Outcome: To Compare the Change in EQ-5D3L Usual Activities Score From Pre-Op to 5 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 5 years
Population: Study terminated early due to slow recruitment rate. 5 Year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

46. Secondary Outcome: To Compare the EQ-5D3L Pain/Discomfort Score Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 3 - 6 months
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 52
Number analyzed (Number of Knees) | 45 | 52
Points | -0.56 (0.81) | -0.67 (0.83)

47. Secondary Outcome: To Compare the EQ-5D3L Pain/Discomfort Score Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 1 year
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 50
Number analyzed (Number of Knees) | 45 | 50
Points | -0.67 (0.77) | -0.68 (0.82)

48. Secondary Outcome: To Compare the EQ-5D3L Pain/Discomfort Score Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 2 years
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 48
Number analyzed (Number of Knees) | 43 | 48
Points | -0.72 (0.83) | -0.60 (0.82)

49. Secondary Outcome: To Compare the Change in EQ-5D3L Pain/Discomfort Score From Pre-Op to 5 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 5 years
Population: Study terminated early due to slow recruitment rate. 5 Year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

50. Secondary Outcome: To Compare the Change in EQ-5D3L Anxiety/Depression Score From Pre-Op to 3 to 6 Months Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 3 - 6 months
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 52
Number analyzed (Number of Knees) | 45 | 52
Points | -0.27 (0.72) | -0.27 (0.63)

51. Secondary Outcome: To Compare the Change in EQ-5D3L Anxiety/Depression Score From Pre-Op to 1 Year Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 1 year
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 50
Number analyzed (Number of Knees) | 45 | 50
Points | -0.24 (0.65) | -0.24 (0.62)

52. Secondary Outcome: To Compare the Change in EQ-5D3L Anxiety/Depression Score From Pre-Op to 2 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 2 years
Population: 106 knees enrolled, 15 of which excluded from analysis due to:{0Deaths + 8 Protocol Violations (4Inv & 4 Contr) + + 4 Revisions (1Inv & 3Contr) + 3 Lost to follow up (2Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 48
Number analyzed (Number of Knees) | 43 | 48
Points | -0.21 (0.80) | -0.17 (0.63)

53. Secondary Outcome: To Compare the Change in EQ-5D3L VAS Score From Pre-Op to 3 to 6 Months Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 3 - 6 months
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 52
Number analyzed (Number of Knees) | 45 | 52
Points | 18.3 (23.7) | 16.4 (23.3)

54. Secondary Outcome: To Compare the Change in EQ-5D3L VAS Score From Pre-Op to 1 Year Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 1 year
Population: 106 knees enrolled, 13 of which excluded from analysis due to:{0Deaths + 8 Protocol Violations (4Inv & 4 Contr) + 2 Lost to follow up (1Inv & 1Contr) + 3 Missing outcome (0Inv & 3Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 45 | 48
Number analyzed (Number of Knees) | 45 | 48
Points | 20.6 (26.5) | 13.6 (26.5)

55. Secondary Outcome: To Compare the Change in EQ-5D3L VAS Score From Pre-Op to 2 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 2 years
Population: 106 knees enrolled, 15 of which excluded from analysis due to:{0Deaths + 8 Protocol Violations (4Inv & 4 Contr) + 4 Revisions (4Inv & 4Contr)+ 3 Lost to follow up (2Inv & 1Contr)}
Measure: Mean (Standard Deviation); unit: Points
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 43 | 48
Number analyzed (Number of Knees) | 43 | 48
Points | 10.8 (24.7) | 11.4 (26.2)

56. Secondary Outcome: To Compare the Change in EQ-5D3L VAS Score From Pre-Op to 5 Years Post-Op Between PFC Sigma RP and PFC Sigma RP-F Treatment Groups.
Description: as for outcome 34
Time Frame: 5 years
Population: Study terminated early due to slow recruitment rate. 5 Year data not available.
Units Other Than Participants: Number of Knees
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Number analyzed (Participants) | 0 | 0
Number analyzed (Number of Knees) | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse event data were collected between treatment time point and 24 month follow up as this study has been terminated early.
Description: Study protocol was designed and executed on using 'knees' as study units. Adverse events were collected based on the knees being investigated, not per participant, it is not possible to regroup data 'per participant'. Therefore the numbers affected and at risk below are referring to knees.
Arm/Group | PFC Sigma RP-F | PFC Sigma RP
Serious Adverse Events (participants affected / at risk) | 7/50 | 7/56
Other Adverse Events (participants affected / at risk) | 0/50 | 0/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PFC Sigma RP-F (N=50) | PFC Sigma RP (N=56)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Joint dislocations (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Pain (General disorders) | 4 (4) | 2 (2)
Allergy to metals (Immune system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
DePuy reserves the right to review the contents of publications in advance.The PI may freely disclose the trial results only after DePuy has been given the opportunity of reviewing the proposed results communications at least 30 days prior to the intended release.DePuy will advise the PI of any perceived errors,omissions or corrections but the PI will retain final editorial control.In case of disagreement,DePuy and the PI will make every effort to meet in order to discuss and resolve any issues.